CLINICAL TRIAL: NCT02640001
Title: Impact of the Introduction in a Heart Surgery ICU of a PCR Technique (Cepheid Xpert® SA Nasal Complete Assay) to Identify Methicillin-sensitive and Methicillin-resistant Staphylococcus Aureus in Nasal and Respiratory Tract Samples
Brief Title: PCR Technique to Identify Methicillin-sensitive and Methicillin-resistant Staphylococcus Aureus in Nasal and Respiratory Tract Samples
Status: Completed | Type: Observational
Sponsor: Emilio Bouza (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Emilio Bouza, Head of Department, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: MICRO.HGUGM-2015-080
Record Dates: First submitted 2015-10-19; First posted 2015-12-28 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2015-07

CONDITIONS: Thoracic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In patients on mechanical ventilation, it is not known whether the identification of S. aureus in LRT samples improves the performance of its nasal detection.

To assess the MSSA or MRSA carrier status of patients requiring mechanical ventilation for more than 48 hours after major heart surgery: comparing the performance of the diagnostic technique Xpert® SA Nasal Complete assay in nasal swab and LRT samples.

DETAILED DESCRIPTION:
Patients undergoing heart surgery require ventilation for more than 48 hours. These patients, placed on mechanical ventilation for a median of 7 days, will be followed weekly until their discharge from hospital. We estimate we will need 500 determinations.

Samples will be obtained according to usual clinical practice. Thus, rather than discarding a sample, it will be subjected to the two laboratory diagnostic techniques (conventional culture and the Xpert® assay). No patient will be subjected to any procedure outside that of routine clinical practice.

Patient with a tracheal tube in whom nasal and LRT secretions can be simultaneously obtained. Patients may also be included if LRT samples can be obtained via a different approach (tracheostomy, fibrobroncoscopy etc.).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years)
* Signed Informed consent
* Patient admitted to the HS-ICU before or after undergoing heart surgery
* Patient on mechanical ventilation for >2 calendar days on the date of event (suspicion of LRT infection) ), taking the day of ventilator placement as day 1
* Patient with a tracheal tube in whom nasal and LRT secretions can be simultaneously obtained. Patients may also be included if LRT samples can be obtained via a different approach (tracheostomy, fibrobroncoscopy etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Heart Surgery-ICU
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Staphylococcus aureus presence in nasal and respiratory tract samples | every 7 days from date of randomization, an average of two weeks
  diagnostic technique Xpert® SA Nasal Complete assay in nasal swab and LRT samples.

CONTACTS AND LOCATIONS:
Locations (1):
- HGU Gregorio Maranon, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Bouza E, Burillo A, de Egea V, Hortal J, Barrio JM, Vicente T, Munoz P, Perez-Granda MJ. Colonization of the nasal airways by Staphylococcus aureus on admission to a major heart surgery operating room: A real-world experience. Enferm Infecc Microbiol Clin (Engl Ed). 2020 Dec;38(10):466-470. doi: 10.1016/j.eimc.2019.07.013. Epub 2019 Oct 23. English, Spanish. PMID 31668380
- [Derived] Bouza E, Burillo A, Munoz P, Valerio M, Barrio JM, Hortal J, Cuerpo G, Perez-Granda MJ. Do lower respiratory tract samples contribute to the assessment of carriage of Staphylococcus aureus in patients undergoing mechanical ventilation after major heart surgery? PLoS One. 2018 Dec 26;13(12):e0207854. doi: 10.1371/journal.pone.0207854. eCollection 2018. PMID 30586363